CLINICAL TRIAL: NCT06835218
Title: PROstate CAncer Real World Evidence Registry: RECURRENT AND METASTATIC PROSTATE CANCER
Brief Title: PROCARE - PROstate Cancer Real World Evidence Registry
Acronym: PROCARE
Status: Recruiting | Type: Observational
Sponsor: UroTrials Company (GmbH) (Network)
Collaborators: Novartis Pharmaceuticals (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: UT-2023-01; U1111-1299-5868 (Registry Identifier: WHO Universal Trial Number); DRKS00033411 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Biochemical Recurrence of Malignant Neoplasm of Prostate; Non-metastatic Castration-resistant Prostate Cancer; Metastatic Hormone-sensitive Prostate Cancer (mHSPC); Metastatic Castration-resistant Prostate Cancer
Keywords: prostate, cancer, metastatic, systemic therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exploratory molecular analyses of leucocyte DNA and RNA, circulating cell-free tumor DNA and RNA (plasma) as well as protein-biomakers (serum) in correlation with clinical outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cohort 1: biochemical recurrence (BCR) after local curative intended treatment
- Cohort 2: non-metastatic castration-resistant prostate cancer (nmCRPC)
- Cohort 3: metastatic hormone-sensitive prostate cancer (mHSPC)
- Cohort 4: metastatic castration-resistant prostate cancer (mCRCP)

SUMMARY:
The aim of this registry study with long-term follow-up is to record the course of therapy and disease in patients with recurrent and metastatic prostate cancer. The following patient groups are planned:

* Patients with a recurrence of PSA after surgical removal or radiation of the prostate due to prostate cancer; so-called PSA recurrence (relapse) or biochemical recurrence.
* Patients with a PSA recurrence who have received treatment by hormone deprivation therapy (so-called androgen deprivation) and in whom the PSA value has nevertheless risen again without spreading to other organs or parts of the body, so-called non-metastatic castration-resistant prostate cancer.
* Patients with proven spread to other organs or parts of the body (= metastases, e.g. in the bone) without hormone deprivation therapy having been initiated, so-called metastatic hormone-sensitive prostate cancer.
* Patients with prostate cancer and spread to other organs or parts of the body (= metastases) in whom the tumor disease has progressed despite hormone withdrawal treatment (e.g. as evidenced by an increase in PSA), so-called metastatic castration-refractory prostate cancer.

These four groups of patients are enrolled and observed independently of each other at different time periods.

DETAILED DESCRIPTION:
This prospective real-world data and long-term follow-up registry study aims at documenting routine treatment and course of disease of patients with metastatic prostate cancer and patients with biochemical recurrence after local treatment. This may include the following patient cohorts:

Cohort 1: biochemical recurrence after local curative intended treatment (e.g. radical prostatectomy, radiotherapy of the prostate or combination thereof) Cohort 2: non-metastatic castration-resistant prostate cancer Cohort 3: metastatic hormone-sensitive prostate cancer Cohort 4: metastatic castration-resistant prostate cancer These cohorts will be recruited independently at various time frames. No specific study treatment is defined. All treatments are prescribed and performed according to each center's medical practice. Any treatment choice or change in regimen is performed at the discretion of each treating physician. During the routine visits, routine data on the course of the disease and therapy are documented for all cohorts at certain time points (after inclusion, then every 3 or 6 months and when changing therapy), standardized quality of life questionnaires (FACT-P and EQ-5D-5L) and biomaterial is collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult prostate cancer patients (age ≥18 years).
* Diagnosis at time of study inclusion Cohort 1: biochemical recurrence (BCR) after local curative intended treatment (e.g. radical prostatectomy, radiotherapy of the prostate or combination thereof) Cohort 2: non-metastatic castration-resistant prostate cancer (nmCRPC) or Cohort 3: metastatic hormone sensitive prostate cancer (mHSPC) or Cohort 4: metastatic castration-resistant prostate cancer (mCRPC) (irrespective of treatment choice, treatment line)
* Patients who will receive a new line of systemic therapy at the time of study entry or up to 4 weeks thereafter. Regarding Cohort 4 this includes patients with a new diagnosis of mCRPC (=first line mCRPC) after either treatment for mHSPC or non-metastatic CRPC as well as patients with prior mCRPC treatments (2nd, 3rd, … line).
* For Cohorts 1, 2 and 3: Disease proven by clinical measures (i.e. standard imaging) to be either unsuitable for local salvage treatment (e.g. surgery, radiotherapy) or local treatment is declined by the patient.
* Patients, who are able and willing to sign the informed consent form

Exclusion Criteria:

• Patients who are not eligible for observation due to severe comorbidities or unavailability according to the treating physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Presence of Prostate
Study Population: Adult prostate cancer patients (age ≥18 years) who will receive a new line of systemic therapy at the time of study entry or up to 4 weeks thereafter.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapy Frequencies and Patterns of Therapy | Through study completion, an average of 7 years
  Description of therapy frequencies and patterns in routine clinical practice for the included patient cohorts

SECONDARY OUTCOMES:
Annual (vs. cumulative) Patterns of Disease Management | Through study completion, an average of 7 years
  Description of annual (vs. cumulative) patterns of disease management i.e. choice of treatment applied in German routine practice (including initial disease/ metastatic diagnosis and previous cancer drug and non-drug treatments)
Methodology for Disease Status Assessment | Through study completion, an average of 7 years
  Methodology used for disease status assessment (e.g. PSA-measurements, imaging)
Frequency for Disease Status Assessment | Through study completion, an average of 7 years
  Frequency for disease status assessment (e.g. PSA-measurements, imaging)
Drug Effectiveness Depending on Prior Treatment | Through study completion, an average of 7 years
  Assessment of drug effectiveness depending on prior use of an ARPI, docetaxel and other drugs in the BCR, nmCRPC and mHSPC setting as well as prior treatments for mCRPC
Parameters Affecting Prognosis | Through study completion, an average of 7 years
  Identification of parameters affecting patients prognosis
Incidence of Adverse Events, serious Adverse Events | Through study completion, an average of 7 years
  Incidence of AEs and sAEs including long term safety and tolerability
Treatment Adherence | Through study completion, an average of 7 years
  Assessment of Treatment Adherence of patients undergoing different treatment regimes within the distinct cohorts
Assessment of Patient Reported Outcomes for cohort 1 | Through study completion, an average of 7 years
  Including Patients Quality of Life affected by Treatment using EORTC QLQ-C30 (cohort 1)
Assessment of Patient Reported Outcomes for cohort 2-4 (EQ-5D-5L) | Through study completion, an average of 7 years
  Including Patients Quality of Life affected by Treatment using EQ-5D-5L
Assessment of Patient Reported Outcomes for cohort 2-4 (FACT-P) | Through study completion, an average of 7 years
  Including Quality of Life by Treatment using FACT-P
Assessment of Patient Paths I | Through study completion, an average of 7 years
  Place of Initial and Metastatic Diagnosis, Involved Treatment Facilities, Tumor Board Decisions
Assessment of Patient Paths II | Through study completion, an average of 7 years
  Type of Initial and Metastatic Diagnosis, Involved Treatment Facilities, Tumor Board Decisions
Applied Imaging Assessments II | Through study completion, an average of 7 years
  PET/CT
Applied Imaging Assessments III | Through study completion, an average of 7 years
  Bone scan
Applied Imaging Assessments IV | Through study completion, an average of 7 years
  PSMA-SPECT/CT
Applied Imaging Assessments V | Through study completion, an average of 7 years
  MRI
Applied Imaging Assessments VI | Through study completion, an average of 7 years
  CT
Applied Imaging Assessments VII | Through study completion, an average of 7 years
  PSMA PET/CT
Description of Patient and Tumor Characteristics | Through study completion, an average of 7 years
  Including Molecular Alterations, if Assessed) in Routine Care of mHSPC and mCRPC Patients

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Oliver Grimm, Professor, Study Director — University Hospital Jena; Boris Hadaschik, Professor, Study Director — University Hospital, Essen
Locations (51):
- Germany (51):
  - National Center for Tumor Dieseases (NCT) Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Hospital Mannheim, Mannheim, Baden-Wurttemberg
  - Medical Office for Urology Nürtingen, Nürtingen, Baden-Wurttemberg
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - University Hospital Augsburg, Augsburg, Bavaria
  - Hospital Bayreuth GmbH, Bayreuth, Bavaria
  - University Hospital Erlangen, Erlangen, Bavaria
  - Hospital Kempten, Kempten (Allgäu), Bavaria
  - Hospital Nürnberg North, Nuremberg, Bavaria
  - Caritas-Hospital St. Josef, Regensburg, Bavaria
  - University Hospital Würzburg, Würzburg, Bavaria
  - "Vivantes Prostatazentrum" Hospital "am Urban", Berlin, Brandenburg
  - University Hospital Hamburg-Eppendorf, Hamburg, Hamburg
  - University Hospital Frankfurt/Main, Frankfurt am Main, Hesse
  - Universitiy Hospital Gießen und Marburg GmbH, Site: Gießen, Giessen, Hesse
  - Universital Hospital Gießen & Marburg GmbH, Site: Marburg, Marburg, Hesse
  - Hospital Wetzlar, Wetzlar, Hesse
  - Medical Office for Urology, Braunschweig, Lower Saxony
  - Medical Office for Urology, Herzberg am Harz, Lower Saxony
  - St. Bernward Hospital Hildesheim, Hildesheim, Lower Saxony
  - St. Bernward Krankenhaus GmbH, Hildesheim, Lower Saxony
  - Medical Office for Urology Altstadtquartier Magdeburg, Magdeburg, Lower Saxony
  - MVZ Onco Medical GmbH Neustadt, Neustadt am Rübenberge, Lower Saxony
  - Praxisgemeinschaft f. Onkologie & Urologie, Wilhelmshaven, Lower Saxony
  - University Hospital Rostock, Rostock, Mecklenburg-Vorpommern
  - University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Medical Office for Urology, Bayenthal, North Rhine-Westphalia
  - Marien Hospital Bergisch Gladbach,, Bergisch Gladbach, North Rhine-Westphalia
  - Johanniter GmbH, Johanniterkrankenhaus, Bonn, North Rhine-Westphalia
  - Johanniter Hosptal Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - Medical Office for Urology "Urologicum", Duisburg, North Rhine-Westphalia
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Marien Hospital Herne, University Hospital der Ruhr-Universität Bochum, Herne, North Rhine-Westphalia
  - "Brüder" Hospital St. Joseph Paderborn, Paderborn, North Rhine-Westphalia
  - University Hospital Wuppertal, Wuppertal, North Rhine-Westphalia
  - Medical Office for Urology, Würselen, North Rhine-Westphalia
  - Urban Hospital Karlsruhe, Karlsruhe, Rhineland-Palatinate
  - Hospital "Barmherzigen Brüder "Trier, Trier, Rhineland-Palatinate
  - Center for Urology Boxberg, Neunkirchen, Saarland
  - University Hospital Leipzig, Leipzig, Saxony
  - City Hospital Dessau, Dessau, Saxony-Anhalt
  - Universitiy Hospital Halle, Halle, Saxony-Anhalt
  - University Hospital Halle, Halle, Saxony-Anhalt
  - Urologie Altstadtquartier Magdeburg, Magdeburg, Saxony-Anhalt
  - University Hospital Magdeburg, Magdeburg, Saxony-Anhalt
  - Univerity Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - University Hospital Jena, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No
A Steering Committee is established for the study. SC will decide about requests for specific analyses. In case of positive opinion analyses will be done in-house and results provided to researchers.